CLINICAL TRIAL: NCT04146519
Title: Developent and Implement a Method of Parkinson's Disease Therapy Using Cell Technology
Brief Title: Parkinson's Disease Therapy Using Cell Technology
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Belarusian Medical Academy of Post-Graduate Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20171292
Record Dates: First submitted 2019-10-18; First posted 2019-10-31 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Transplantation:Mesenchymal Stem Cell Transplantation
Keywords: Parkinson's disease; mesenchymal stem cells; intranasal transplantation; intravenous transplantation; tandem transplantation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Autologous MMSC
  Interventions: Biological: Autologous mesenchymal stem cells
- control group (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Autologous mesenchymal stem cells — Autologous mesenchymal stem cells
  Arms: Study group
Other: Placebo — Saline solution
  Arms: control group

SUMMARY:
Treatment of patients with Parkinson's disease using mesenchymal stem cells is a perspective method to influence on the pathogenesis of the disease. At the same time, this is a complex and still insufficiently explored process. Autologous mesenchymal stem cells will be transplanted to 30 patients with Parkinson's disease. The results of the effectiveness of the combined and intravenous routes of mesenchymal stem cells administration on the motor and non-motor symptoms in these patients will be evaluated and compared with the results of control group that received placebo therapy

ELIGIBILITY:
Inclusion Criteria:

1. A reliable diagnosis of Parkinson's disease, according to the diagnostic criteria developed by the Brain Bank of the Society for Parkinson's disease of Great Britain (UK Brain Bank Criteria, 1992).
2. Stage of the disease according to Hen-Yar: 1.5 - 3.0 stage.
3. Rapidly progressive type with a change in the stages of Parkinson's disease in no more than 4 years.
4. A good response to levodopa treatment: a positive dopamine test for assessing motor functions by a total score of section 3 of the UPDRS scale in the on- and off-period (not less than 30%).
5. The duration of the disease is not more than 8 years with the absence of motor fluctuations and dyskinesias.
6. The age of patients is up to 65 years

Exclusion Criteria:

e and parkinsonism-plus. 2. Severe concomitant diseases (congestive heart failure, myocardial infarction, pneumonia, decompensated diabetes mellitus, cachexia, etc.).

3. Autoimmune diseases, a tendency to bleeding, a history of sepsis. 4. Oncological diseases. 5. The presence of acute or exacerbation of the chronic inflammatory process of the sinuses or oral cavity.

6. A positive result for HIV, hepatitis B (HBV), hepatitis C (HCV), syphilis (RW).

7. Cognitive deficit. 8. Mental disorders - hallucinations, behavior disorders. 9. Depression of a pronounced degree (not more than 19 points on the Hamilton scale).

10. Alcoholism, drug addiction, criminal liability in the patient's history. 11. Pregnancy, lactation.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
motor symptoms change | 3 month
  Positive trend is going to be detected in the overall score of the third part of the UPDRS scale(Unified Parkinson Disease Rating Scale) in the off- and in the on-period:neurological examination of patients in the dynamics is carried out in the morning after a 12 (24) - hour break in taking anti-Parkinsonian drugs "off-state", then one hour after they were taken "on-state".
  A score of 64 on the third part of the UPDRS scale represents the worst (total motor disability) with a score of zero representing (no disability).
non-motor symptoms change | 3 month
  Identification and assessment of the severity of non-motor symptoms is carried out using Non-motor Symptoms Questionnaire (PD NMS Questionnaire).A score of 30 represents the worst result with a score of zero representing (no disability).
sleep quality change | 3 month
  The Pittsburgh Sleep Quality Index (PSQI) is used to assess sleep quality over the last month.The sleep component scores are summed to yield a total score ranging from 0 to 21 with the higher total score (referred to as global score) indicating worse sleep quality.
daytime sleepiness change | 3 month
  The Epworth Sleepiness Scale (ESS) is used to measure daytime sleepiness.The ESS score can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity in daily life (ASP), or their 'daytime sleepiness'.
signs of depression change | 3 month
  We use the Hamilton Depression Scale - Hamilton psychiatric rating scale for depression (HDRS) - to identify signs of depression. A score of 52 represents the worst result with a score of zero representing (no disability).

CONTACTS AND LOCATIONS:
Locations (1):
- the Belarusian Medical Academy of Postgraduate Education, Minsk, Belarus

REFERENCES:
- [Background] Boika A, Aleinikava N, Chyzhyk V, Zafranskaya M, Nizheharodava D, Ponomarev V. Mesenchymal stem cells in Parkinson's disease: Motor and nonmotor symptoms in the early posttransplant period. Surg Neurol Int. 2020 Nov 11;11:380. doi: 10.25259/SNI_233_2020. eCollection 2020. PMID 33408914